CLINICAL TRIAL: NCT06199141
Title: The Impact of Multi-drug Resistant Gram-negative Bacteria on Outcomes in Patients Requiring Veno-venous Extracorporeal Membrane Oxygenation (ECMO)
Brief Title: Multi-drug Resistant Gram-negative Bacteria and Veno-venous Extracorporeal Membrane Oxygenation (ECMO)
Acronym: MDR-ECMO
Status: Completed | Type: Observational
Sponsor: University of Padova (Other)
Collaborators: Azienda Ospedaliera Mater Domini di Catanzaro (Unknown); Policlinico di Bari Giovanni XXIII (Unknown); Azienda Ospedaliera Universitaria Integrata Verona (Other); Fondazione IRCCS San Gerardo di Monza (Unknown)
Responsible Party: Principal Investigator, Annalisa Boscolo, Co-investigator, University of Padova
Other Study IDs: MDR GN bacteria in VV-ECMO
Record Dates: First submitted 2023-12-26; First posted 2024-01-10 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Respiratory Distress Syndrome, Adult; Multi-antibiotic Resistance
Keywords: ARDS; Multi-antibiotic Resistance; extracorporeal membrane oxygenation
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- VV-ECMO patients: Patients requiring VV-ECMO for acute respiratory distress syndrome (ARDS)

SUMMARY:
Veno-venous extracorporeal membrane oxygenation (VV-ECMO) is a life-support technique used in patients with most severe acute respiratory distress syndrome (ARDS). ARDS is a life-threatening form of respiratory failure associated with a mortality rate of approximately 40-45%.Despite several studies confirming a real benefit of the use of ECMO in patients with ARDS who are unresponsive to conventional management, ECMO is still a complex and costly treatment that can be exposed to potential complications, such as nosocomial infections (NI).

DETAILED DESCRIPTION:
Noteworthy, the most frequent NIs occurring during VV-ECMO are pneumonia (>40%) and, secondly, blood-stream infections (3-18%). The situation is more challenging for Gram-negative bacilli: more than one-half of the Escherichia coli and more than one-third of the Klebsiella pneumoniae isolates were resistant to at least one antimicrobial group. Of note, an alarming increase in carbapenem resistance has been reported in several species, including K. pneumoniae (7.9% of isolates), P.aeruginosa (16.5% of isolates) and A. baumannii (>30% of isolates).

In fact, the isolation of MDROs has been shown to be an independent risk of death and of subsequent infections not only in critically ill patients but also in those patients requiring VV-ECMO (mortality rate between 56-68%). However, data are still conflicting about the exact incidence of multidrug resistant organisms (MDRO) during VV-ECMO and the impact on short- and mid-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* ARDS
* VV-ECMO

Exclusion Criteria:

* pregnancy
* age < 18
* uncompleted records
* survival < 24h after ECMO connection

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients affected by ARDS (according to Berlon criteria) undergoing VV-ECMO.
Sampling Method: Probability Sample
Enrollment: 279 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Overall incidence of MDR Gram negative bacteria isolations | From ECMO connection up to 48 hours after ECMO de-connection
  Overall incidence of MDR Gram negative bacteria isolations during ECMO (n° events/1.000 person-days of ECMO)
Incidence of MDR Gram negative bacteria acquired | From ECMO connection up to 48 hours after ECMO de-connection
  Incidence of MDR Gram negative bacteria acquired after ECMO connection (n° events/1.000 person-days of ECMO)
Incidence of MDR Gram negative bacteria isolated prior to ECMO connection | At study enrollment
  Incidence of patients requiring VV-ECMO with a previous MDR Gram negative bacteria

SECONDARY OUTCOMES:
Incidence of MDR-related infections (plus descriptive analysis) | From ECMO connection up to 48 hours after ECMO de-connection
  Incidence of patients acquiring MDR-related infections
Incidence of MDR-related colonizations (plus descriptive analysis) | From ECMO connection up to 48 hours after ECMO de-connection
  Incidence of patients acquiring MDR-related colonizations
Risk factors-mortality | At ECMO connection (baseline)
  Risk factors for mortality

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Bruni, Prof, Principal Investigator — Azienda Ospedaliera Mater Domini di Catanzaro
Locations (1):
- Azienda Ospedaliera Università Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boscolo A, Bruni A, Giani M, Garofalo E, Sella N, Pettenuzzo T, Bombino M, Palcani M, Rezoagli E, Pozzi M, Falcioni E, Pistollato E, Biamonte E, Murgolo F, D'Arrigo G, Gori M, Tripepi GL, Gottin L, Longhini F, Grasso S, Navalesi P, Foti G. Retrospective ANalysis of multi-drug resistant Gram-nEgative bacteRia on veno-venous extracorporeal membrane oxygenation. The multicenter RANGER STUDY. Crit Care. 2024 Aug 27;28(1):279. doi: 10.1186/s13054-024-05068-x. PMID 39192287